CLINICAL TRIAL: NCT02103101
Title: Influence of ABCB1 Polymorphisms on Plasma Concentrations of New Oral Anticoagulants in Case of Serious Adverse Events
Acronym: Pgp NACO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Etablissement Français du Sang (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pgp NOAC
Record Dates: First submitted 2014-03-31; First posted 2014-04-03 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Anticoagulants; Thromboembolism; Hemorrhage
Keywords: polymorphism; ABCB1; P-glycoprotein; oral anticoagulant; dabigatran; apixaban; rivaroxaban; hemorrhagic complication; thrombo-embolism; serious adverse event
MeSH Terms: conditions — Thromboembolism; Hemorrhage | interventions — ATP Binding Cassette Transporter, Subfamily B, Member 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study cohort (Other): Measurement of Plasma Concentrations of NOACs Identification of ABCB1 polymorphisms coding for P-gp
  All patients aged over 18 and less than 80 years admitted for a serious adverse event (bleeding or thrombo-embolic complication) while under treatment with any of the following oral anticoagulant agents: dabigatran, rivaroxaban or apixaban. Blood samples will be drawn to measure plasma concentrations of the oral anticoagulant agent at the time of the adverse event, and presence of polymorphisms of ABCB1 will be investigated.
  Interventions: Other: Measurement of Plasma Concentrations of NOACs; Genetic: Identification of ABCB1 polymorphisms coding for P-gp

INTERVENTIONS:
Other: Measurement of Plasma Concentrations of NOACs — Plasma concentrations of dabigatran, rivaroxaban or apixaban will be measured using High Performance Liquid Chromatography (HPLC) coupled with tandem mass spectrometry (MS/MS). Blood samples will be taken in an EDTA tube and rapidly centrifugated. Plasma will be aliquoted and frozen at minus 80 degrees Celsius for later analysis.
Genetic: Identification of ABCB1 polymorphisms coding for P-gp — To investigate the existence of a relation between polymorphisms of ABCB1 and plasma concentrations of new oral anticoagulants, the SNaPshot® Multiplex System will be used enabling multiplexing of SNPs (single nucleotide polymorphisms) of the ABCB1 gene (namely rs4148738, rs2235046, rs1128503, rs10276036, rs1202169, rs1202168, rs1202167).

SUMMARY:
Vitamin K antagonists were hampered by several disadvantages, such as the need for frequent monitoring. In this context, new oral anticoagulants (NOACs) have been developed and are now available on the market. These NOACs, like all anticoagulant drugs, continue to be associated with an increased risk of bleeding. In addition, the lack of antidote and the absence of valid data regarding biological monitoring can pose problems in case of overdose or when emergency surgery is required. Studies investigating the pharmacokinetic properties of rivaroxaban and dabigatran, two NOACs now approved for the market, have shown high variability between individuals, with coefficients of variation of up to 60% for some pharmacokinetic parameters in patients treated after orthopaedic surgery. The relation between plasma concentrations of NOAC and bleeding risk has been clearly established in clinical trials.

Dabigtran, rivaroxaban and apixaban are known substrates of P-glycoprotein (Pgp). Pgp activity can be affected by pharmacological inducing or inhibiting agents. This can lead to a significant change in the pharmacokinetics of NOACs, with a decrease or increase (respectively) in the level of intestinal absorption, leading to respectively reduced or increased plasma concentrations of the drug. Furthermore, there exist genetic mutations of Pgp, presenting in particular a lower level of activity than the non-mutated protein. We hypothesized that the polymorphisms (mutations) of the ABCB1 gene that codes for Pgp could influence plasma concentrations of dabigatran, rivaroxaban and apixaban, and consequently, impact on the concentration of NOACs and as a corollary, on the bleeding and thromboembolic risk of patients treated with these molecules.

The main objective of this study is to study the relation between polymorphisms of the ABCB1 gene that codes for Pgp and plasma concentrations of NOACs in patients treated for a hemorrhagic or thromboembolic complication occurring under NOAC therapy.

Secondary objectives are to evaluate the distribution of ABCB1 polymorphisms among the various hemorrhagic risk factors, and to compare the frequency of the polymorphism in patients from the study population vs the general population.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >18 and <80 years of age
* Patients admitted to the University Hospital of Besancon for a serious adverse event (major bleeding complication or thrombo-embolic event) occurring under treatment with any one of the three commercially available new oral anticoagulant agents (rivaroxaban, apixaban or dabigatran).
* Patients must have social security coverage.
* Patients must provide written informed consent.

Exclusion Criteria:

* Hemorrhagic complication from causes not related to drug therapy
* Hemorrhagic complication occurring in patients not treated with oral anticoagulants at the time of the event
* Thrombo-embolic complication occurring in patients not treated with oral anticoagulants at the time of the event
* Legal incapacity, patients under judicial protection
* Patients with no social security coverage
* Patients unlikely to be compliant or anticipated by the investigator to be non-compliant with the study requirements
* Patients in a wash-out period further to participation in a previous clinical trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2014-11-13 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Measurement of plasma concentrations of new oral anticoagulant agents | 0 days (at inclusion)
  Plasma concentrations of dabigatran, rivaroxaban or apixaban will be measured using High Performance Liquid Chromatography (HPLC) coupled with tandem mass spectrometry (MS/MS). Blood samples will be taken in an EDTA tube and rapidly centrifugated. Plasma will be aliquoted and frozen at minus 80 degrees Celsius for later analysis.
Identification of polymorphisms of the gene ABCB1 coding for P-gp | 0 days (at inclusion)
  To investigate the existence of a relation between polymorphisms of ABCB1 and plasma concentrations of new oral anticoagulants, the SNaPshot® Multiplex System will be used enabling multiplexing of SNPs (single nucleotide polymorphisms) of the ABCB1 gene (namely rs4148738, rs2235046, rs1128503, rs10276036, rs1202169, rs1202168, rs1202167).

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas F Meneveau, MD, PhD, Principal Investigator — Centre Hospitalier Universitaire de Besancon
Locations (1):
- CHU Besancon, Besançon, France